CLINICAL TRIAL: NCT01131104
Title: A Prospective Case-crossover Study to Evaluate the Possible Association Between the Use of PDE5 Inhibitors and the Risk of Acute Nonarteritic Anterior Ischemic Optic Neuropathy (NAION)
Brief Title: A Study to Determine if There is a Possible Association Between NAION and Phosphodiesterase Type 5 (PDE5) Inhibitors
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 11638; H6D-MC-LVHQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-10; First posted 2010-05-26 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2017-09

CONDITIONS: Nonarteritic Anterior Ischemic Optic Neuropathy
Keywords: NAION
MeSH Terms: conditions — Optic Neuropathy, Ischemic | interventions — Phosphodiesterase 5 Inhibitors; Tadalafil; Sildenafil Citrate; Vardenafil Dihydrochloride

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with NAION who have used PDE5 inhibitors
  Interventions: Drug: PDE5 Inhibitors

INTERVENTIONS:
Drug: PDE5 Inhibitors — Observational study of participants who have been prescribed phosphodiesterase type 5 (PDE5) inhibitors by their physician during routine clinical practice.
  Other Names: tadalafil; sildenafil; vardenafil

SUMMARY:
Study H6D-MC-LVHQ is an observational, non-interventional, multi-center, prospective, case-crossover study to evaluate the possible association between the use of phosphodiesterase type 5 (PDE5) inhibitors and the risk of acute nonarteritic anterior ischemic optic neuropathy (NAION) in males. Subjects with newly diagnosed NAION will be asked via a structured questionnaire about their use of PDE5 inhibitors and other risk factors prior to the onset of their vision loss.

ELIGIBILITY:
Inclusion Criteria:

* Adult male subjects, at least 18 years of age, who are willing to participate in the study
* Participants who experienced abrupt visual loss in one eye (defined as typically less than a 1-day period or visual loss noted upon awakening) and presented for an initial visit within 45 days of onset of NAION symptoms to an ophthalmologist that resulted in a diagnosis of Suspected NAION by the investigator

Exclusion Criteria:

* Previous history of NAION
* Previous history of arteritis (anywhere in the body) or clinical or diagnostic testing evidence of temporal arteritis
* History of glaucoma in either one or both eyes
* History of multiple sclerosis or diagnostic testing evidence of optic neuritis
* Have dementia or other reasons for memory impairment in the opinion of the investigator
* Have participated in other non-observational studies within 3 months of NAION onset

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential cases of acute NAION will be prospectively identified by approximately 20 neuro-ophthalmology centers in the US
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2010-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fr- 9 AM-5 PM Eastern time (UTC?GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (44):
- United States (44):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Cockerham Eye Consultant, Los Altos, California
  - Precision Eye Care, National City, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Russell P Edwards M.D., San Diego, California
  - Pacific Eye Associates, San Francisco, California
  - Eye Surgical & Medical Associates, Inc., Visalia, California
  - The Eye Care Group, New Haven, Connecticut
  - Avail Clinical Research LLC, DeLand, Florida
  - University of Florida - Gainesville, Gainesville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - USF Eye Institute, Tampa, Florida
  - University of Illinois At Chicago Med Center, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Northshore Eye and Vision Center, Glenview, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Univ KY Clinical Resch Org- KY Clinic, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Bethesda Neurology, LLC, Bethesda, Maryland
  - Longwood Medical Eye Center, Boston, Massachusetts
  - Atlantic Clinical Trials, LLC, Watertown, Massachusetts
  - Henry Ford Health System, Dearborn, Michigan
  - Neuro-Ophthalmic Services, Royal Oak, Michigan
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - JFK Medical Center, NJ Neuroscience Institute, Edison, New Jersey
  - Stony Brook University Medical Center, East Setauket, New York
  - E.S. Harkness Eye Institute, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Ohio State Univ College Of Medicine, Columbus, Ohio
  - Dr. Daniel Lin, Oregon, Ohio
  - Family Eye Care, Lancaster, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Allegheny Ophthalmic & Orbital Associates, Pittsburgh, Pennsylvania
  - Retina Consultants of Charleston, Charleston, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Neuro-Opthalmology of Texas, Houston, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington
  - Swedish Neuroscience Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Set were enrolled participants who met inclusion/exclusion criteria and physician-diagnosed Nonarteritic Anterior Ischemic Optic Neuropathy (NAION)known date of onset.
  Adjudication-Confirmed NAION Set were confirmed participants (by adjudication committee) with inclusion/exclusion criteria and physician-diagnosed NAION known date of onset.
Groups:
- Enrolled Set: Enrolled participants who met inclusion/exclusion criteria and had physician-diagnosed NAION with a known date of onset.
Period: Overall Study
Arm/Group | Enrolled Set
Started | 345
Study Set | 344
Adjudication-Confirmed NAION Set | 279
30-Day Analysis Set (Participants had adjudication-confirmed NAION and complete PDE5 inhibitor information.) | 24
42-Day Analysis Set (Participants had adjudication-confirmed NAION and complete PDE5 inhibitor information.) | 28
12-Month Analysis Set (Participants had adjudication-confirmed NAION and complete PDE5 inhibitor information.) | 26
Completed | 332
Not Completed | 13
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 4
Not completed — Information Not Available | 5
Not completed — No Information on Index Date of Onset | 1

BASELINE CHARACTERISTICS:
Population: Participants with adjudication-confirmed NAION.
Arm/Group | Cohort 1
Number analyzed (Participants) | 279
Age, Customized [Mean (Standard Deviation); unit: years] | 61.5 (10.70)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 0
  Male | 279
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  Caucasian | 267
  More than one race | 2
  Unknown or Not Reported | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 265
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 279
Adjudicated NAION Participants within the 30-Day Analysis Set [Count of Participants; unit: Participants] | 24

OUTCOME MEASURES:

1. Primary Outcome: 30-Day Person Time Analysis Risk of NAION Associated With PDE5 Inhibitor Use
Description: Total participant days of PDE5 inhibitor exposure within 30 days prior to onset of NAION.
Time Frame: 30 days prior to NAION onset
Population: All participants in the 30 day analysis set.
Measure: Number (95% Confidence Interval); unit: Relative risk of exposure
Units Other Than Participants: Participant days
Arm/Group | Cohort 1
Number analyzed (Participants) | 24
Number analyzed (Participant days) | 720
Relative risk of exposure | 2.27 [0.99 to 5.20]

ADVERSE EVENTS:
Description: No serious adverse events or other adverse events were assessed or collected, with the exception of NAION.
Arm/Group | Cohort 1
Serious Adverse Events (participants affected / at risk) | 0/345
Other Adverse Events (participants affected / at risk) | 0/345

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days